CLINICAL TRIAL: NCT00703105
Title: Defining the Role of CD4+CD25+ Immunoregulatory T-cells in the Treatment of Patients With Advanced Ovarian Cancer Who Receive Dendritic Cell Based Vaccine Therapies
Brief Title: Ovarian Dendritic Cell Vaccine Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Patrick Stiff, Professor of Medicine, Director, Cardinal Bernardin Cancer Center, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200541
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; Tregs; vaccine; Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Dendritic Cell Vaccination (Experimental): DC vaccination with 1 x 10(6th) tumor lysate or WT1 and MUC1 peptide and KLH-loaded immature DCs into inguinal nodes identified by ultrasound guidance for a total of three injections at two week intervals(6 weeks)
  Interventions: Biological: DC vaccination

INTERVENTIONS:
Biological: DC vaccination — DC vaccination with 1 x 10(6th) tumor lysate or tumor peptides and KLH-loaded immature DCs into inguinal nodes identified by ultrasound guidance for a total of three injections at two week intervals; (6 weeks)

SUMMARY:
The purpose of this study is to determine if a dendritic cell vaccine made with autologous tumor lysate or for patients who are HLA-A2 with peptides of MUC1 and WT1 therapy will produce remissions in patients with advanced ovarian cancer. This research is being done because we want to find new therapies for treatment of relapsed or refractory (resistant to ordinary treatment) ovarian cancer. The use of vaccine therapy is research.

A new experimental approach for treating refractory or relapsed ovarian cancer involves using the patients own immune system to kill the cancer cells. These immune cells are called monocytes and are harvested from blood. The process of Leukapheresis collects the monocytes called Dendritic Cells. This is usually a 3 hour process done in the comfort of a hospital bed in the apheresis lab, similar to giving blood for donation. Approximately 300cc's are collected during this process, the equivalent of about 10 ounces of blood. Once these dendritic cells are collected - a special laboratory grows and processes them into a vaccine using a patient's own tumor cells or for those with a specific HLA type (HLA-A2) with tumor peptides. This preparation is then given back to the patient hopefully to stimulate the immune system to kill cancer cells. This type of treatment is considered biological research.

DETAILED DESCRIPTION:
Patients with advanced ovarian carcinoma who have failed initial curative chemotherapy attempts will be evaluated at the time of relapse for tumor debulking surgery prior to the initiation of salvage chemotherapy. If appropriate, samples will be collected for tumor lysate preparation for vaccination as per the existing Loyola protocol. Lysates may also be produced by the collection of malignant effusions as performed for palliation of symptoms. Patients will then receive palliative chemotherapy to a maximum tumor cytoreduction. Patients from whom sufficient tumor cells have been collected for DC-based vaccine production will undergo a leukapheresis for DC cell production. Once completed, these patients will receive a DC vaccination with 1 x 106 tumor lysate and KLH-loaded immature DCs into inguinal nodes identified by ultrasound guidance for a total of three injections at two week intervals; or for those who are HLA-A2 restricted with pharmaceutical grade MUC1 and WT1 tumor peptides.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic or cytologic diagnosis of epithelial ovarian cancer
* Patients are eligible if they have failed to enter a complete remission after therapy and are not eligible for otherwise curative therapy
* Patients must not have received any antineoplastic chemotherapy or immunotherapy for the four weeks preceding tumor excision; six weeks for nitrosoureas and mitomycin-C
* Patients must not have received irradiation for the four weeks prior to removal of the tumor and no previously irradiated tumor deposits may be used for tumor lysate in the development of the dendritic cell vaccine
* Age >18 years. Because no dosing or adverse event data are currently available on the use of dendritic cell vaccination in patients <18 years of age, children are excluded from this study but may be eligible for future pediatric phase 2 combination trials
* Life expectancy of greater than three months
* Karnofsky performance status must be >70%; (see appendix A)
* Patients must have adequate baseline hematopoetic function as defined below. - The following labs must be drawn within four weeks of having the tumor harvested and/or receiving the vaccine

  * total white blood cell count > 2,500/mm3
  * absolute neutrophil count > 1,000/mm3
  * absolute lymphocyte count > 500/mm3
  * platelet count > 80,000/mm3
* Patients must have adequate baseline organ function as defined below. The following labs must be drawn within four weeks of having the tumor harvested and/or receiving the vaccine:

  * total bilirubin ≤ 2.0 mg/dl
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine ≤2.0 mg/dl
  * prothrombin time (INR) ≤1.5 X institutional upper limit of normal
  * albumin >3.0 mg/dl
* If patients have had recent surgery, then they must be fully recovered from the effects of that surgery.
* The effects of the vaccine on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Additional eligibility requirements for vaccine therapy initiation:

* Patients are eligible after tumor collection for the vaccine strategy, or for those selected to receive ONTAK alone (group 3 -CLOSED) because tumor is not available can enroll at ay time they fulfill the Eligibility Criteria. Pre-vaccination the goal is to establish a Minimal Residual Disease state (MRD maximum tumor diameter of any residual disease ≤ 1cm). This can be achieved with surgery and/or salvage chemotherapy. Vaccine administration and/or vaccine therapy will commence at least 4 weeks after the completion of the last day of any of the aforementioned therapies
* Patients to be randomized to groups 1 and 2 must have tumor available for preparation of tumor lysate vaccine
* Women and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents.
* Patients who have received prior anti-tumor vaccines are ineligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to monocolonal antibodies from Murine sources
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active bleeding, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled bronchospasm, hypertension, hyperglycemia, or hypercalcemia; or psychiatric illness/social situations that in the opinion of the investigators would compromise the patient's ability to tolerate this treatment or affect compliance
* Pregnant and lactating women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants, breastfeeding should be discontinued if the mother is treated with the vaccine. These potential risks may also apply to other agents used in this study
* Patients with HIV infection, AIDS, or hepatitis B surface antigen positivity, are excluded from this trial. Patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* History of corticosteroid use in the four weeks preceding entry onto the clinical trial, or the requirement for ongoing corticosteroid use during the study period
* Patients who are expected to require therapeutic anticoagulation during the trial period
* Patients with known brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-10; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
To determine if administration of an autologous tumor lysate or tumor peptide-loaded dendritic cell vaccine enhances the immune response in patients with relapsed/refractory ovarian cancer | days 45 and 62 post vaccine
  response rate

SECONDARY OUTCOMES:
To characterize the toxicities of this novel DC-based vaccination strategy. | weekly assessments for a total of 4 weeks
  CTAE4 toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stiff, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola Univeristy Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois, United States